CLINICAL TRIAL: NCT05006300
Title: Evaluation of the Efficacy and Tolerance of Topialyse Baume Barriere in Children With Atopic Dermatitis: Randomised, Multicentric, Open-label Study
Brief Title: Evaluation of the Efficacy of Topialyse Baume barrière on Atopic Dermatis
Acronym: TOPIA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment long and complicated
Sponsor: SVR Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOPIA-2021.03; 2021-A00613-38 (Other: French Agency for the Safety of Health Products (ANSM))
Record Dates: First submitted 2021-08-03; First posted 2021-08-16 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): One application of Topialyse Baume Barrière per day
  Interventions: Other: Topialyse Baume Barrière
- Group 2 (Experimental): Two applications of Topialyse Baume Barrière per day
  Interventions: Other: Topialyse Baume Barrière

INTERVENTIONS:
Other: Topialyse Baume Barrière — Evaluation of the efficacy of the cosmetic product SVR TOPIALYSE Baume Barrière on the reduction of topical corticosteroid consumption in children from 3 months to 17 years old presenting mild to moderate atopic dermatitis after 28 and 56 days of use, at one or two apllications /day.

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of a new SVR care product and to evaluate the reduction of the topical corticosteroids' consumption with this emollient care.

Atopic dermatitis is a vicious circle that must be broken, but certain aggravating factors are added to this circle. There is a lot of talk about pollution but, more recently, studies have been carried out on the worsening role of dust mites on atopic skin.

The SVR product is therefore based on it:

TOPIALYSE Baume Barrière is a care product that is lipid-replenishing, repairing and protective: a triple reinforced action for 48 hours: anti-scratching, anti-irritation, and anti-external aggression.

DETAILED DESCRIPTION:
1. RATIONALE

The mainstay of treatment for Atopic dermatitis (AD) is use of emollient and topical medications. Topical corticosteroids are the gold standard of anti-inflammatory therapy in AD especially AD flare-ups, in order to reduce inflammation and pruritus. Their long-term use is associated with the risk of local and systemic adverse effects.

The purpose of this study is to evaluate the efficacy and tolerability of TOPIALYSE Baume Barrière and to evaluate the reduction of the topical corticosteroids' consumption with this emollient care.

2 STUDY OBJECTIVES

2.1 PRIMARY OBJECTIVE: The main objective of this study is to evaluate the efficacy of the cosmetic product SVR TOPIALYSE Baume Barrière on the reduction of topical corticosteroid consumption in children from 3 months to 17 years old presenting mild to moderate atopic dermatitis (5 < SCORAD < 40), after 28 days of use.

2.2 SECONDARY OBJECTIVE: 2.2.1. To evaluate the efficacy of the study product after 28 and 56 days of use on children of 3 months to 17 years with mild to moderate atopic dermatitis by the following criteria:

1. Number of flare-up
2. SCORAD
3. Amount of topical corticosteroid consumption
4. Mean PO-SCORAD
5. Quality of life
6. Skin condition and functional skin signs

   2.2.2 Evaluate the tolerance of the study product after 28 and 56 days of use on children 3 months to 17 years old with mild to moderate atopic dermatitis

   2.2.3. To evaluate the persistent effect of the cosmetic product SVR TOPIALYSE Barrier Balm after 24 and 48 hours of stopping use on children from 3 months to 17 years old with mild to moderate atopic dermatitis

   3 STUDY METHODOLOGY This is a multicentric, randomized and open-label study. It is an interventional study with minimal risks (Category 2).

   3.1 EVALUATION CRITERIA (see outcomes part)

   3.2 EVALUATION METHODS

   3.2.1 Topical corticosteroid consumption Consumption of class 2 or 3 topical corticosteroids will be assessed throughout the study by the number of days of use and the weight of the topical corticosteroid tube per month.

   3.2.2 SCORAD At D -37, D -7, D0, D28 and D56, the dermatologist calculates the objective SCORAD over the entire body.

   A. First, the investigator assesses the distribution of atopic dermatitis by calculating the extent. For each zone, the investigator evaluates the proportion of the zone considered affected by atopic dermatitis compared to the suggested maximum score.

   B. Second, the investigator scores the intensity of the following parameters: erythema, oedema/papules, oozing/crust, excoriation, lichenification and xerosis

   C. Finally, the investigator questions the subjects about their subjective symptoms: pruritus abd insomnia

   The total score of the objective SCORAD is obtained according to the following formula:

   SCORAD = A/5 + 7 B/2 + C

   3.2.3 Skin condition assessment 3.2.4 IDQOL questionnaire 3.2.5 Local tolerance assessment 3.2.6 Cutaneous functional signs assessment 3.2.7 Study product questionnaire 3.2.8 Standardized photographs

   4 SELECTION OF STUDY POPULATION Sixty-two children (62) will be enrolled in the study. The subjects will be recruited via the Necker Volunteer Database or from those who spontaneously come to the Necker Children's Hospital or the Pr. Tennstedt' medical office or if needed, via press advertising after approval by the Ethics Committee.

   5. DURATION OF TREATMENT, DOSING AND ADMINISTRATION 5.1 Duration of treatment Depending on the group, the tested products will be applied for fifty-six days either consecutively (Group 1) or with one application every two days (Group 2).

   6 INVESTIGATIONAL PLAN 6.1 STUDY DESIGN This is a multicentric, randomized and open-label study. It is an interventional study with minimal risks (Category 2).

   The study will be performed in 62 children with mild to moderate atopic dermatitis. The screening of the subjects will be performed at the Necker-Enfants malades hospital and at the Pr Tennstedt medical office within three weeks (D -58) prior to the enrollment visit at D -37 and to allow verification of the subject compatibility with the inclusion and exclusion criteria.

   6.1.1 Study location The study will be performed in two Investigation centers, the Necker-Enfant malades hospital, authorized by the Regional Agency of Health (ARS) to perform biomedical research and the Pr. Tennstedt medical office.

   6.1.2 Study duration The study participation for each subject will last up to 3 months (21 days for screening and 95 days of clinical participation).

   6.2 STUDY PROCEDURES

   6.2.1 Screening visit (visit 1): D -58 to D -37 The screening visit will be performed within three weeks of the day before D -37. The following procedures may be carried on several days if needed.
   * Subject information and presentation of the informed consent form,
   * Inclusion/ exclusion criteria checking. 6.2.2 Enrollment/ inclusion visit (Visit 2), phase 1: D -37

   The subject will have to come to the investigator site for:
   * Inclusion/ exclusion criteria checking,
   * Informed consent signature,
   * Medical history and concomitant therapies,
   * Physical examination: general aspects, height, weight,
   * Vital signs: sitting systolic and diastolic blood pressure (mm-Hg) and pulse rate (beats per minute) after a 5-minute rest,
   * Clinical scoring with the SCORAD (Scoring Atopic Dermatitis),
   * Recording information on the topical corticosteroid usually used in the atopic dermatitis flare-up on the source file and the e-CRF,
   * Weighing and recording the weight of the topical corticosteroid tube on the source folder and the e-CRF,
   * Distribution of patient diary for adverse events and number of relapses,
   * Distribution of patient cards with study information,
   * Downloading of the PO-SCORAD (Patient-Oriented Scoring Atopic Dermatitis) mobile application by the subjects' parents and explanation of the instructions and dates for filling in the booklet,
   * Evaluation of the quality of life with IDQOL (Infant's Dermatitis Quality of Life index) questionnaire,
   * Standardized photographs if desired and authorized,
   * Appointment for the next visits on D-7, D0, D28, D56, D57 and D58 and record them on the patient diary and patient study card.
   * Provision of the patient diary.

   Between this visit and the next:
   * Use of the usual emollient,
   * Application of the usual topical corticosteroid in case of atopic dermatitis flare-up,
   * Weekly filling of the PO-SCORAD,
   * Filling of the patient diary every day.

   6.2.3 Follow-up visit 1 (visit 3), end of phase 1: D -7
   * Checking the patient diary,
   * Verification of adverse events,
   * Verification of concomitant medication modifications,
   * Weighing and recording the weight of the topical corticosteroid tube on the source folder and the e-CRF,
   * Completion of the source files and the e-CRF,
   * Subject is randomized according to a randomization list (attributed in chronological order),
   * Dermatological examination by local 5-point tolerance scale by the investigator,
   * SCORAD clinical scoring,
   * Evaluation of the quality of life with IDQOL (Infant's Dermatitis Quality of Life Index) questionnaire,
   * Standardized photographs if desired and authorized,
   * Reminder of the next D0 appointment.

   6.2.4 Wash-out period: D-7 to D0 After this visit, the patients have to stop using the usual emollient and the usual topical corticosteroid, weekly filling of the PO-SCORAD application and filling out the patient diary every day.

   6.2.5 Follow up visit 2 (visit 4), starting phase 2: D0
   * Checking the patient diary,
   * Verification of adverse events,
   * Verification of concomitant medication modifications,
   * Completion of the source files and the e-CRF,
   * SCORAD clinical scoring,
   * Dermatological examination by local 5-point tolerance scale by the investigator or co-investigator,
   * Scoring of skin condition by the investigator or co-investigator,
   * Assessment questionnaire of skin condition by the subject' parent,
   * Assessment questionnaire of tolerance and signs of skin intolerance by the subject' parent,
   * ID-QOL questionnaire,
   * Standardized photographs if desired and authorized
   * Product distribution,
   * Weighing of study products and topical corticosteroid recording in the source folder and e-CRF,
   * First pat of the product,
   * Reminder of the next T28 appointment.

   Between this visit and the next:
   * Use of the TOPIALYSE emollient once a day or once every 2 days depending on randomization,
   * Application of the usual topical corticosteroid in case of atopic dermatitis flare-up,
   * Weekly filling of the PO-SCORAD,
   * Filling of the patient diary every day.

   6.2.6 Follow-up visit 3 (Visit 5), phase 2: D28

   - Checking the patient diary,
   * Verification of adverse events,
   * Verification of concomitant medication modifications,
   * Completion of the source files and the e-CRF,
   * SCORAD clinical scoring,
   * Dermatological examination by local 5-point tolerance scale by the investigator or co-investigator,
   * Scoring of skin condition by the investigator or co-investigator,
   * Assessment questionnaire of skin condition by the subject' parent,
   * Assessment questionnaire of tolerance and signs of skin intolerance by the subject' parent,
   * ID-QOL questionnaire,
   * Standardized photographs if desired and authorized,
   * Weighing of study products and topical corticosteroid recording in the source folder and e-CRF,
   * Reminder of the next T56 appointment.

   Between this visit and the next:

   - Use of the TOPIALYSE emollient once a day or once every 2 days depending on randomization,
   * Application of the usual topical corticosteroid in case of atopic dermatitis flare-up,
   * Weekly filling of the PO-SCORAD,
   * Filling of the patient diary every day.

   6.2.7 Follow-up visit 4 (visit 6), phase 2: D56

   - Checking the patient diary,
   * Verification of adverse events,
   * Verification of concomitant medication modifications,
   * Completion of the source files and the e-CRF,
   * SCORAD clinical scoring,
   * Dermatological examination by local 5-point tolerance scale by the investigator or co-investigator,
   * Scoring of skin condition by the investigator or co-investigator,
   * Assessment questionnaire of skin conditions by the subject' parent,
   * Assessment questionnaire of tolerance and signs of skin intolerance by the subject' parent,
   * ID-QOL questionnaire,
   * Subjective assessment questionnaire on the study product by the subject' parent,
   * Standardized photographs if desired and authorized,
   * Weighing of study products and topical corticosteroid recording in the source folder and e-CRF,
   * Collection of the patient diary,
   * Collection of study products.

   After this visit, the patients have to stop using the TOPIALYSE Baume Barrière emollient and the topical corticosteroid.

   6.2.8 Follow-up visit 5, phase 2: D57 - Assessment questionnaire for skin condition,
   * Questionnaire for assessment of tolerance and signs of skin intolerance,
   * Filling the PO-SCORAD. This part will only be done by the subject' parent and send to the study center.

   6.2.9 Follow-up visit 6/ End of Study: D58 - Assessment questionnaire for skin condition,

   - Questionnaire for assessment of tolerance and signs of skin intolerance,

   - Filling the PO-SCORAD,

   - Delivery of documents to the investigator centre. This part will only be done by the subject' parent and send to the study center.

   7 STATISTICAL METHODS 7.1 BASELINE CHARACTERISTICS Continuous demographic variables (e.g. age, weight, and height) will be summarized, using mean, standard deviation, minimum, maximum and number of available observations.

   Qualitative demographic characteristics will be summarized by counts and percent. Other subject characteristics (anomalies in physical examination, prior medication, inclusion / exclusion checklist) will be listed only.

   7.2 STATISTICAL ANALYSES Descriptive statistics (N, mean, standard error, min, max,) will be calculated by test product for each parameter.

   Prior to any statistical analysis, the normality of each variable will be tested using the Shapiro Wilks test of normality.

   Statistical Tests:

   For each normal variable, comparisons will be performed using a t-test for paired data.

   For each non normal variable, comparison will be performed using a Wilcoxon rank sum test.

   7.3 NUMBER OF SUBJECTS CALCULATION In the treatment of atopic dermatitis, the use of a simple emollient makes it possible to reduce by about 10% the amount of topical corticosteroid used [33]. In the present study, it is expected that TOPIALYSE Baume Barrière applied 1 application/day will reduce the consumption of topical corticosteroid by at least 35% after 28 days of application based on the results of the study of GIORDANO-LABADIE et al, 2006. Calculation of the number of patients by the Arcsinus method shows that 31 patients would allow to detect a significant difference between TOPIALYSE Baume Barrière applied 1 application/day and the reference value 10% with a power of 95% at risk α =0.05 (bilateral test). It is also expected that TOPIALYSE Baume Barrière applied 1 application/2 days will lead to a comparable decrease, therefore 31 patients will also be included in this group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 3 months and 17 years old;
2. Female or male subjects;
3. Subjects of Caucasian origin with skin type I to IV according to the Fitzpatrick scale
4. Subject with atopic background and mild to moderate signs of atopic dermatitis on the face and/or the body - 5<SCORAD<40 [2] - with or without dust mite sensitivity;
5. Subject who had at least one atopic dermatitis flare-up in the month prior to the study;
6. Subject with dry to very dry skin on the face and the body;
7. Subject who used a topical corticosteroid - class 2 or 3 - during a flare-up in the month prior to the study;
8. Subject regularly using an emollient in the management of atopic dermatitis;
9. Subject agreeing not to expose to sunlight or artificial UV rays during the study period;
10. Subject who, in the Investigator's opinion, will comply with the requirements of the protocol (e.g., follow protocol instructions, have regular contact to allow evaluation during the study);
11. Subject agreeing not to use any other facial or body care product during the study period, except study products and their usual emollient;
12. Subject agreeing not to use any face or body care products 24 hours prior to the start of the study;
13. Subject agreeing not to use hygiene products with a moisturizing, nourishing, or anti-drying effect during the study period and at least 24 hours before the start of the study;
14. Subject agreeing not to carry out an oral corticosteroid treatment during the entire study period;
15. Patients whose legal guardian has given written consent for their participation in the study;
16. Subject related to the Social Security of a parent or legal guardian in agreement with the French law on interventional research.

Exclusion Criteria:

1. Subject has known or suspected allergies or sensitivities to any of the constituents of the test product (see Product labels);
2. Subject has a medical condition or is taking medication that could put him or her at undue risk;
3. Subject has an unstable medical condition or one that could interfere with the study;
4. Subject who has not received any topical corticosteroids in the month prior to the start of the study;
5. Subject who received oral corticosteroids during the three months before the start of the study;
6. Subject who received oral immunosuppressive drugs during the three months prior to the start of the study;
7. Subject who received local immunosuppressants during the month prior to the start of the study;
8. Subject who received antihistamines during the week prior to the start of the study;
9. Subject having an underlying known disease, or surgical, physical, or medical condition that, in the opinion of the Investigator might interfere with the interpretation of the clinical trial results such as:

   * History of other recurrent dermatologic conditions (e.g., psoriasis, eczema, urticarial, and/or hives);
   * Any systemic, local disease or skin condition (i.e., active cutaneous diseases; scars, moles, excessive hair, non-flat area, sunburn, uneven skin coloration or other blemishes) on the body;
10. Subject is currently receiving treatment that may interfere, in the opinion of the Investigator, with interpretation of the study results;
11. Subjects taking part in another study or being excluded from a previous study.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the topical corticosteroid consumption with the use of Topialyse Baume Barrière (1month) | DAY 28
  Evaluation of the reduce of amount of topical corticosteroid by comparing the number of days of use and the weight of class 2 or 3 topical corticosteroid per month before and after the use of the cosmetic product (TOPIALYSE Baume Barrière)

SECONDARY OUTCOMES:
Evaluation of the topical corticosteroid consumption with the use of Topialyse Baume Barrière (1month) | DAY 56
  Evaluation of the effectiveness of the cosmetic product (TOPIALYSE Baume Barrière) on the reduction of the quantity of topical corticosteroid by comparing the number of days of use and the weight of class 2 or 3 topical corticosteroid per month at D56 versus D -7.
Evaluation of the efficacy of the product by reducing the number of atopic dermatitis flare-ups | DAY 28 and DAY 56
  Evaluation of the efficacy of the product by reducing the number of atopic dermatitis flare-ups per month at D28 and D56 versus D0.
Evaluation of the efficacy of the product by reducing the SCORAD (Scoring of Atopic Dermatitis) | DAY 28 and DAY 56
  Evaluation of the efficacy of the product by reducing the SCORAD (Scoring of Atopic Dermatitis) (Appendix n°1) at D28 and D56 versus D0 and versus D -7 and D -37.
Evaluation of the product's effectiveness by reduction of the mean PO-SCORAD (Patient Oriented Scoring of Atopic Dermatitis) per month | DAY 28, DAY 56, DAY 57 and DAY 58
  Evaluation of the product's effectiveness by reduction of the mean PO-SCORAD (Patient Oriented Scoring of Atopic Dermatitis) (Appendix n°2) per month at D28, D56, D57 and D58 versus D0.
Evaluation of the efficacy of the product on the skin condition by a dermatologist on a 5-point scale. | DAY 28 and DAY 56
  Evaluation of the efficacy of the product on the skin condition (Appendix n°3) by a dermatologist on a 5-point scale (0 to 4) at D28 and D56 versus D0.
Evaluation of the efficacy of the product on the cutaneous condition. | DAY 28, DAY 56, DAY 57 and DAY 58
  Evaluation of the efficacy of the product on the cutaneous condition (nourished and moisturized aspect of the skin) by a self-evaluation or carried out by the volunteer's parent on a 5-point scale (0 to 4) at D28, D56, D57 and D58 versus D0.
Evaluation of the effect of the product on the improvement of the quality of life of children | DAY 28 and DAY 56
  Evaluation of the effect of the product on the improvement of the quality of life of children using the IDQOL (Infant's Dermatitis Quality Of Life index) questionnaire (Appendix n°4) at D28 and D56 versus D0.

IPD SHARING:
Plan to Share IPD: No